CLINICAL TRIAL: NCT03652688
Title: Group-based Intervention for Alcohol, Drugs and Aggression Among Club Patrons
Brief Title: Group-based Intervention for Club Patrons
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Pacific Institute for Research and Evaluation (Other)
Collaborators: Klein Buendel, Inc. (Industry)
Responsible Party: Principal Investigator, Brenda Miller, Senior Scientist, Pacific Institute for Research and Evaluation
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AA022331
Record Dates: First submitted 2018-04-16; First posted 2018-08-29 (Actual); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2025-01

CONDITIONS: Drink Too Much; Drinking, Binge; Drunk; Drug Use; Aggression; Aggression Sexual; Peer Group; Safety Issues; Harm Reduction
Keywords: nightclubs; bars; alcohol; drugs; aggression; harm reduction
MeSH Terms: conditions — Binge Drinking; Alcoholic Intoxication; Aggression; Harm Reduction

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Participant
Masking Description: Groups assigned to experimental and control conditions were given a tablet on which either the experimental or control program was provided. Both groups were told that they would be viewing a program on safety while at the club. Both groups had to respond to some questions on the tablet about the program. Both groups were asked to interact as a group to answer these questions. Without a view of the tablet, it appeared as if both experimental and controls had the same condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nightlife Safety Plans (NSP) (Experimental): Observed indicators that a group member may be in trouble due identified risks were provided and if detected, they were given practical skills on implementing the 3 0's: Outreach, Options, and Out. Outreach consisted of techniques for approaching your friend and acquiring more information whether there was a problem. Options were to be employed if problems were confirmed and were designed to provide easy, simple steps to reduce risks and decrease probability of escalation of problems. Out refers to the plans the group made before entering the club that they would leave as a group to keep the group members safe. Group commitment to implement these safety steps was emphasized. Interactive and visually attractive scenes were drawn as graphic images to avoid didactic delivery.
  Interventions: Behavioral: Nightlife Safety Plans (NSP)
- Fire Safety (Sham Comparator): Groups in the control condition were also given information on safety and the focus of this safety message was regarding fires in nightclubs. Groups were given didactic materials to read with some still images. There were a few questions for the group to address.
  Interventions: Behavioral: Fire Safety

INTERVENTIONS:
Behavioral: Nightlife Safety Plans (NSP) — A group approach to reducing unwanted outcomes was implemented prior to entering the nightclub. The focus was on peer-to-peer intervention.
  Arms: Nightlife Safety Plans (NSP)
Behavioral: Fire Safety — Groups were asked to read information about fire safety prior to entering the club and to answer some questions about fire safety
  Arms: Fire Safety

SUMMARY:
The purpose of this study is to develop and test a group-based strategy for encouraging groups of young adults who are engaged in party behaviors at nightclubs to intervene with each other to reduce harms associated with overuse of alcohol and recreational drugs and to reduce harms associated with aggression (physical and sexual).

DETAILED DESCRIPTION:
This study focuses on high risk behaviors (excessive alcohol use, drug use) and unwanted experiences (physical/sexual aggression) that may occur during an evening at a night club for young adults engaged in party behaviors. the goals were: 1) to develop a screener that accurately assesses a group's level of risk for one specific night of club attendance and based upon this assessment, (2) to provide naturally occurring social groups with the necessary skills to identify vulnerability for and to provide them with tools to reduce harms. An algorithm calculated in real time during an entrance survey predicted the types of risks that the group members may encounter during the evening based upon past behaviors and expectations for the evening. Social groups in the experimental condition were exposed to a brief intervention that focused on developing skills described as the 3 O's: a) Outreach-how to approach fellow group members who are at risk, (b) Options-how to suggest options that would increase safety and (c) Out-How to assess when it is time to leave the club. This brief, interactive intervention was delivered by small tablet computers that utilized mobile application technology and cellular wireless service. This low cost delivery was considered important to providing later adoption in the real world and the interactive nature of the intervention was designed to appeal to the young adult population.

ELIGIBILITY:
Inclusion Criteria:

* Must be within age range, entering the club that night, group size must be 2 or more

Exclusion Criteria:

* working or performing at the club that night

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 959 (Actual)
Dates: Start 2016-06-15 (Actual); Primary Completion 2017-10-01 (Actual); Study Completion 2017-10-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brenda A Miller, Ph.D., Principal Investigator — Pacific Institute for Research and Evaluation
Locations (2):
- United States (2):
  - Brenda Miller, Berkeley, California
  - Prevention Research Center, Berkeley, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Byrnes HF, Miller BA, Bourdeau B, Johnson MB. Impact of Group Cohesion Among Drinking Groups at Nightclubs on Risk From Alcohol and Other Drug Use. J Drug Issues. 2019 Oct;49(4):668-679. doi: 10.1177/0022042619859257. Epub 2019 Sep 8. PMID 34658404
- [Result] Byrnes HF, Miller BA, Bourdeau B, Johnson MB, Buller DB, Berteletti J, Rogers VA. Prevention of Alcohol and Other Drug Overuse Among Nightclub Patrons: A Randomized Trial of a Group-Based Mobile Intervention at Nightclubs. J Stud Alcohol Drugs. 2019 Jul;80(4):423-430. doi: 10.15288/jsad.2019.80.423. PMID 31495379

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Individuals who arrived in Groups (2+ people) were recruited as they were entering the club. Not everyone in the group had to agree to participate to be eligible. No names were collected at recruitment.
Pre-assignment Details: Individuals who arrived in Groups (2+ people) were recruited as they were entering the club. Not everyone in the group had to agree to participate to be eligible. No names were collected at recruitment.
Units Other Than Participants: groups
Groups:
- Nightlife Safety Plans: Observed indicators that an individual may be in trouble due identified risks were provided and if detected, they were given practical skills on implementing the 3 0's: Outreach, Options, and Out. Outreach consisted of techniques for approaching your friend and acquiring more information whether there was a problem. Options were to be employed if problems were confirmed and were designed to provide easy, simple steps to reduce risks and decrease probability of escalation of problems. Out refers to the plans the peer group made before entering the club that they would leave as a group to keep each other safe. Commitment to implement these safety steps was emphasized. Interactive and visually attractive scenes were drawn as graphic images to avoid didactic delivery.
  Three 0's: A peer approach to reducing unwanted outcomes was implemented prior to entering the nightclub. The focus was on peer-to-peer intervention.
- Fire Safety: Individuals in the control condition were also given information on safety and the focus of this safety message was regarding fires in nightclubs. They were given didactic materials to read with some still images. There were a few questions for the peer group to address.
  Fire Safety: They were asked to read information about fire safety prior to entering the club and to answer some questions about fire safety
Period: Baseline
Arm/Group | Nightlife Safety Plans | Fire Safety
Started | 459; 173 groups | 500; 179 groups
Completed | 459; 173 groups | 497; 179 groups
Not Completed | 0; 0 groups | 3; 0 groups
Not completed — Withdrawal by Subject | 0 | 3
Period: Follow-up
Arm/Group | Nightlife Safety Plans | Fire Safety
Started | 459; 173 groups | 497; 179 groups (Although enrolled, only 497 completed the control condition)
Completed | 403; 156 groups | 443; 164 groups
Not Completed | 56; 17 groups | 54; 15 groups
Not completed — Lost to Follow-up | 56 | 54

BASELINE CHARACTERISTICS:
Groups:
- Nightlife Safety Plans (NSP): Observed indicators that a group member may be in trouble due identified risks were provided and if detected, they were given practical skills on implementing the 3 0's: Outreach, Options, and Out. Outreach consisted of techniques for approaching your friend and acquiring more information whether there was a problem. Options were to be employed if problems were confirmed and were designed to provide easy, simple steps to reduce risks and decrease probability of escalation of problems. Out refers to the plans the group made before entering the club that they would leave as a group to keep the group members safe. Group commitment to implement these safety steps was emphasized. Interactive and visually attractive scenes were drawn as graphic images to avoid didactic delivery.
  Three 0's: A group approach to reducing unwanted outcomes was implemented prior to entering the nightclub. The focus was on peer-to-peer intervention.
- Total: Total of all reporting groups
Arm/Group | Nightlife Safety Plans (NSP) | Fire Safety | Total
Number analyzed (Participants) | 459 | 500 | 959
Age, Continuous [Mean (Standard Deviation); unit: years] | 27.63 (6.10) | 28.31 (6.56) | 27.99 (6.35)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female | 195 | 218 | 413
  male | 247 | 255 | 502
  transgender woman | 1 | 2 | 3
  transgender male | 1 | 0 | 1
  refused/unidentified | 15 | 25 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 97 | 93 | 190
  Not Hispanic or Latino | 334 | 375 | 709
  Unknown or Not Reported | 28 | 32 | 60
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 6 | 12
  Asian | 88 | 115 | 203
  Native Hawaiian or Other Pacific Islander | 10 | 6 | 16
  Black or African American | 28 | 47 | 75
  White | 205 | 213 | 418
  More than one race | 39 | 28 | 67
  Unknown or Not Reported | 83 | 85 | 168
Region of Enrollment [Number; unit: participants]
  United States | 459 | 500 | 959
Legally intoxicated by alcohol [Count of Participants; unit: Participants] — Breath tests using a breathalyzer that resulted in a percent of alcohol in breath that was .05% or higher was considered evidence of alcohol impairment or intoxication. Population: Breath tests to determine the level of alcohol use was not obtained on all participants due to equipment or recording failure.
  Participants
    number analyzed (Participants) | 436 | 479 | 915
    (all) | 105 | 151 | 256

OUTCOME MEASURES:

1. Primary Outcome: Number of Safety Actions Taken to Intervene Within Group
Description: Five types of safety actions were assessed for individuals (as they exited the club) that could have occurred in response to peer's use of alcohol or drugs, experiencing physical aggression and/or sexual aggression. These safety actions were: (1) checked in with friends to assess their safety, (2) monitored alcohol consumption of peers, (3) encouraged peer to pace their drinking, (4) discouraged drug use, and (5) encouraged steps to sober up. An individual could report 0-5 safety actions. Because this was a peer group intervention, a mean score was created for each group by adding the total individual scores within each group, (groups ranged in size from 2-9, making this total possible range 0-45) and dividing these total within group scores by the number in the group. Thus, each peer group had a score ranging from 0-5, with the higher the score, the more protective the group was.
Time Frame: On average, follow up data was collected 1 hour and 54 minutes after baseline (SD 1 hour 3 minutes). The range was from 9 minutes to 5 hours and 15 minutes.
Population: The number of cases analyzed is less than the total number who returned for follow-up due to incomplete exit surveys.
Measure: Mean (Standard Deviation); unit: score on a scale
Units Other Than Participants: groups
Arm/Group | Nightlife Safety Plans (NSP) | Fire Safety
Number analyzed (Participants) | 372 | 433
Number analyzed (groups) | 173 | 179
score on a scale | 2.14 (0.96) | 1.90 (0.85)
Statistical Analysis 1: Comparison: Nightlife Safety Plans (NSP) vs Fire Safety; The unit of analyses was the individual, nested within groups; Test type: Superiority; p < 0.001, ANOVA; F = 14.463

2. Primary Outcome: Protective Action Reported for Physical Aggression Incident
Description: Among those who experienced physical aggression, the prevalence of a group member taking action(s) to intervene was reported.
Time Frame: as for outcome 1
Population: Only individuals who had experienced physical aggression could possibly have someone take action to intervene, hence the overall number of participants analyzed is smaller.
Measure: Count of Participants; unit: Participants
Groups:
- Nightlife Safety Plans: Observed indicators that a group member may be in trouble due identified risks were provided and if detected, they were given practical skills on implementing the 3 0's: Outreach, Options, and Out. Outreach consisted of techniques for approaching your friend and acquiring more information whether there was a problem. Options were to be employed if problems were confirmed and were designed to provide easy, simple steps to reduce risks and decrease probability of escalation of problems. Out refers to the plans the group made before entering the club that they would leave as a group to keep the group members safe. Group commitment to implement these safety steps was emphasized. Interactive and visually attractive scenes were drawn as graphic images to avoid didactic delivery.
  Three 0's: A group approach to reducing unwanted outcomes was implemented prior to entering the nightclub. The focus was on peer-to-peer intervention.
Arm/Group | Nightlife Safety Plans | Fire Safety
Number analyzed (Participants) | 45 | 34
Participants | 9 | 3
Statistical Analysis 1: Comparison: Nightlife Safety Plans vs Fire Safety; Test type: Superiority; p = .08, Chi-squared, Corrected

3. Primary Outcome: Protective Action Reported for Sexual Aggression Incident
Description: Among those who experienced sexual aggression, the prevalence of a group member taking action(s) to intervene was reported.
Time Frame: as for outcome 1
Population: Analyses based upon those who reported an incident of sexual aggression as those who had not experienced sexual aggression would not have received any safety actions from a group member.
Measure: Count of Participants; unit: Participants
Arm/Group | Nightlife Safety Plans | Fire Safety
Number analyzed (Participants) | 45 | 34
Participants | 16 | 11
Statistical Analysis 1: Comparison: Nightlife Safety Plans vs Fire Safety; Test type: Superiority; p = 0.954, Chi-squared, Corrected

4. Secondary Outcome: Legally Intoxicated
Description: Percent who were legally intoxicated (BAC.08% or higher)
Time Frame: as for outcome 1
Population: Legal intoxication was determined by the use of a breath test. The discrepancy between the overall number of participants included at follow-up was lower due to equipment (breathalyzer) data was unable to be linked to a specific person either due to equipment malfunction or human error.
Measure: Count of Participants; unit: Participants
Arm/Group | Nightlife Safety Plans | Fire Safety
Number analyzed (Participants) | 390 | 429
Participants | 151 | 189
Statistical Analysis 1: Comparison: Nightlife Safety Plans vs Fire Safety; Test type: Superiority; p = .035, Chi-squared, Corrected; Chi-Square = 4.436

5. Secondary Outcome: Prevalence of Recreational Drug Use
Description: Any use of recreational drugs present in oral fluid tests based upon lab results
Time Frame: as for outcome 1
Population: The population analyzed is smaller than the number or respondents who completed follow-up due to refusals to give oral fluid samples for analyses or human error resulting in inability to link the oral fluid sample with a specific person.
Measure: Count of Participants; unit: Participants
Arm/Group | Nightlife Safety Plans | Fire Safety
Number analyzed (Participants) | 393 | 435
Participants | 141 | 132
Statistical Analysis 1: Comparison: Nightlife Safety Plans vs Fire Safety; Test type: Superiority; p = .106, Chi-squared, Corrected; Chi-Square = 2.615

6. Secondary Outcome: Leaving Club With Friend(s) Arrived With
Description: Prevalence of safety action to leave club with friends that arrived with
Time Frame: as for outcome 1
Population: Missing data accounts for the lower number of cases in each of the conditions due to not completing the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Nightlife Safety Plans | Fire Safety
Number analyzed (Participants) | 393 | 435
Participants | 345 | 342
Statistical Analysis 1: Comparison: Nightlife Safety Plans vs Fire Safety; Test type: Superiority; p < 0.001, Chi-squared, Corrected; Chi-Square = 11.636

7. Other Pre Specified Outcome: Experienced Physical Aggression
Description: While at the club, someone intentionally pushed, shoved, or punched the respondent
Time Frame: as for outcome 1
Population: The number of cases analyzed is less than the total number who returned for follow-up due to incomplete exit surveys and non-response to item.
Measure: Count of Participants; unit: Participants
Arm/Group | Nightlife Safety Plans | Fire Safety
Number analyzed (Participants) | 362 | 406
Participants | 37 | 39

8. Other Pre Specified Outcome: Experienced Sexual Aggression
Description: While at the club, the respondent experienced someone touching them sexually in a way that they did not want to be touched or did something else sexual to the respondent that they did not want them to do
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Nightlife Safety Plans | Fire Safety
Number analyzed (Participants) | 376 | 410
Participants | 52 | 40

9. Other Pre Specified Outcome: Sexual Harassment
Description: Respondent experienced someone sexually coming on to person after indicating no interest
Time Frame: as for outcome 1
Population: as for outcome 7
Measure: Count of Participants; unit: Participants
Arm/Group | Nightlife Safety Plans | Fire Safety
Number analyzed (Participants) | 375 | 408
Participants | 50 | 52

ADVERSE EVENTS:
Time Frame: On average, follow up data was collected 1 hour and 54 minutes after baseline (SD 1 hour 3 minutes). The range was from 9 minutes to 5 hours and 15 minutes.
Arm/Group | Nightlife Safety Plans (NSP) | Fire Safety
All-Cause Mortality (participants affected / at risk) | 0/459 | 0/500
Serious Adverse Events (participants affected / at risk) | 0/459 | 0/500
Other Adverse Events (participants affected / at risk) | 0/459 | 0/500

LIMITATIONS AND CAVEATS:
Trials were conducted in San Francisco Bay Area thus represent one geographical location

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-01-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT03652688/Prot_SAP_000.pdf
  • Informed Consent Form (2014-01-09): https://cdn.clinicaltrials.gov/large-docs/88/NCT03652688/ICF_001.pdf